CLINICAL TRIAL: NCT07220850
Title: Testing a Multi-behavioral Intervention to Improve Oral Health Behaviors in the Pediatric Dental Surgery Population
Brief Title: Oral Health Intervention for Caregivers of Children Presenting for Dental Surgery
Acronym: PROTECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Helen Lee, MPI, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UH3DE032003 (NIH); UH3DE032003 (NIH)
Record Dates: First submitted 2025-10-21; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Early Childhood Caries
Keywords: Early Childhood Caries; Behavioral Intervention; Community Health Workers
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care: Control (No Intervention): The control, or Usual Care (UC) group will receive usual clinical care, which consists of education during and immediately after surgery. Families randomized to the UC arm will receive the usual standard of care between the time they are identified as surgical candidates to the point when they are scheduled to have their post-surgical visit. Clinical education is provided by pediatric dental residents, and at least one pre-surgical visit is designed to allow families to discuss how their oral health behaviors contribute to caries and answer any questions regarding changing oral health behaviors. Families who are experiencing significant social issues which interfere with their ability to care for their child's teeth are identified by clinic staff and referred to a full-time social worker employed by the dental clinic. Similar to the intervention arm participants, RAs will be trained to report any potential social issues to the research team's clinical psychologist for referral.
- PROTECT Arm: This is the behavioral intervention arm (Experimental): PROTECT (Preventing Recurrent Operations Targeting Early Childhood Caries Treatment) is a 6-month parenting program using evidence-based strategies to increase children's toothbrushing and reduce sugar intake. Sessions also address positive parenting, goal setting, stress management, and problem-solving. Community health workers (CHWs)-some bilingual in Spanish-will deliver 10 sessions (5 informational, 5 maintenance) to caregivers of children scheduled for dental surgery at UIC. Each 30-60-minute session focuses on applying skills to daily life and overcoming behavior-change challenges. CHWs can connect caregivers to social services or dental providers and refer concerns to a clinic social worker through a clinical psychologist. The program, developed from prior evidence and oral health/CHW curricula, covers oral health, nutrition, parenting, rewards, routines, problem-solving, monitoring, self-efficacy, and goal setting.
  Interventions: Behavioral: Behavioral Treatment

INTERVENTIONS:
Behavioral: Behavioral Treatment — PROTECT (Preventing Recurrent Operations Targeting Early Childhood Caries Treatment) is a 6-month parenting program using evidence-based strategies to increase children's toothbrushing and reduce sugar intake. Sessions also address positive parenting, goal setting, stress management, and problem-solving. Community health workers (CHWs)-some bilingual in Spanish-will deliver 10 sessions (5 informational, 5 maintenance) to caregivers of children scheduled for dental surgery at UIC. Each 30-60-minute session focuses on applying skills to daily life and overcoming behavior-change challenges. CHWs can connect caregivers to social services or dental providers and refer concerns to a clinic social worker through a clinical psychologist. The program, developed from prior evidence and oral health/CHW curricula, covers oral health, nutrition, parenting, rewards, routines, problem-solving, monitoring, self-efficacy, and goal setting.
  Arms: PROTECT Arm: This is the behavioral intervention arm

SUMMARY:
Too many young children, particularly those living in poverty, present for dental surgery under anesthesia - an expensive, potentially dangerous, short-term fix that often results in recurring oral health disease and subsequent surgeries. Dr. Helen Lee, an anesthesiologist, and Dr. Joanna Buscemi, a clinical health psychologist, recognized that to decrease need for surgeries, caregivers need resources and support to build their skills and knowledge around managing their child's oral health. After 5 years of relationship-building, publishing preliminary qualitative work, and building a team with the appropriate skills and knowledge, they developed a grant application to develop and test a parenting intervention for caregivers of preschool- aged children presenting for dental surgery.

With support from the National Institute of Dental and Craniofacial Research (NIDCR) of the National Institutes of Health (NIH), the team created the PROTECT intervention with a focus on providing caregivers with parenting and behavioral tools to help improve tooth brushing and lower added sugar intake while simultaneously addressing social determinants of health that make behavior change more difficult. Community health workers will engage with caregivers for 6 months following the child's surgery to deliver PROTECT and support parents in behavioral change. A surgical event is a unique opportunity to change behaviors in systemically oppressed families that have manifested a need for behavior change. This intervention will meet caregivers needs at a critical time when risk disease recurrence intersects with a desire to change. This work has the potential to not only improve oral health of entire households but may also have a concomitant effect on parallel diseases, such as pediatric obesity.

DETAILED DESCRIPTION:
Dental caries is the most common chronic disease of childhood, disproportionately affecting vulnerable children (ethnic/racial minority groups, low-income families, and those who live in rural areas). Young children who have poor oral health behaviors (e.g., inadequate tooth brushing, diet high in added sugar) are at risk for developing severe early childhood caries (S-ECC), which is an indication for dental surgery. Prevalence of S-ECC has declined and utilization of preventive dental care has increased over time. However, inequities in disease burden persist, and demand for dental surgery under general anesthesia (DGA) is increasing. The impact of S-ECC on a child's health ripples out across systemic and psychosocial well-being, with links to childhood obesity and oral health quality of life. Surgical events have inherent safety risks with the potential for iatrogenic errors or possible direct harm. Further, surgical intervention is expensive and ineffective in the long term. Because the intervention does not directly address the etiologic factors, which are largely behavioral, approximately 50% of children have recurrent disease within 12 months after DGA.

Given that parenting behaviors influence a child's oral health status, caregivers are an important catalyst for promoting child behavior changes. Positive parenting, such as appropriate monitoring of a child during tooth brushing or negotiating conflicts when children want sugary snacks, influences child health behaviors. Our team conducted preliminary qualitative research with caregivers while their child was undergoing DGA. This preliminary work, as well as other supportive studies, identified barriers to changing oral health behaviors: parenting style, dental self-efficacy, and oral health knowledge. The objective of this study is to develop and test the initial efficacy of PROTECT (Preventing Recurrent Operations Targeting Early Childhood Caries Treatment), a 6-month behavioral parenting intervention for DGA families enrolled in Medicaid. Our primary outcomes (tooth brushing frequency and % total calories from added sugar) are associated with S-ECC and have been identified as predominant behavior challenges for surgical families. PROTECT, informed by Social Cognitive Theory (SCT), will be delivered by trained community health workers (CHWs) who have social proximity to our participants. PROTECT will be delivered over a six-month interval beginning at the surgical event. This time period coincides with when many parents report high motivation to change behaviors and improve oral health. Behavioral parenting interventions have been validated in mental health and childhood obesity, and we believe will impact S-ECC.

UG3 Specific Aim 1. Develop PROTECT, a 6-month behavioral parenting intervention to reduce S-ECC. The development of PROTECT will be informed by evidence-based behavioral parenting and dietary interventions for preschool children of low-income as well as stakeholder (caregiver, clinical provider, CHW) input.

UG3 Specific Aim 2. Assess the feasibility and accessibility of PROTECT during the perioperative period. We will identify barriers to recruitment, retention, intervention delivery, and outcome measurements. We will recruit 25 caregivers of preschool children scheduled for DGA to conduct a 6-month pilot study with the following goals: finalize study protocol; measure intervention adherence (dose delivered/dose intended); and determine how to optimize intervention via (1) total intervention duration; (2) frequency; and (3) intensity. We will also assess feasibility and acceptability using validated measures.31 UH3 Specific Aim 1. Test the efficacy of PROTECT compared to Usual Care (UC), to improve behavioral oral health outcomes. We will conduct a randomized clinical trial to test the efficacy of PROTECT (n = 210) compared to UC (n = 210) in the pediatric DGA population. Primary outcomes include tooth brushing frequency and % total calories derived from added sugars. We hypothesize that participants in the PROTECT group will increase tooth brushing and decrease % added sugar intake to a greater degree than those in the UC group. Assessments will occur throughout the 6-month intervention and 6 months after intervention completion.

Aim 1a. Determine mechanistic role of behavioral change targets in influencing intervention effectiveness. Per SCT, we will estimate a mediation model with positive parenting, self-efficacy and knowledge as mediators in the pathway to behavioral change. We will also collect weekly remote assessment data (parenting and oral health behaviors), via a text messaging platform, to measure in-the-moment parental behaviors and barriers to adhering to study goals around child oral health behaviors.

A surgical event is a unique opportunity to change behaviors in systemically oppressed families that have manifested a need for behavior change. This proposal will meet caregivers needs at a critical time when risk disease recurrence intersects with a desire to change. This work has the potential to not only improve oral health of entire households but may also have a concomitant effect on parallel diseases, such as pediatric obesity.

ELIGIBILITY:
Inclusion Criteria:

* caregivers of child patients who are in the same household greater than or equal to 50% of the week
* caregivers aged 18-90 years
* caregivers with access to a computer or a telephone
* child patients that are less than 96 months of age at the time of enrollment scheduled for DGA at the UIC clinic

Exclusion Criteria:

* surgical child is foster status
* families who are planning to move out of state within the six-month period
* children with systemic health issues as classified by American Society of Anesthesiology Classification of greater than or equal to 3, or a mental health condition such as autism/developmental delay, as medical complexity is associated with other issues that influence a child's health behaviors and caregiver-child interactions
* and adults unable to consent.

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Basic Research Factors Questionnaire (BRFQ) | 12 months; from baseline to 12 months post-surgical event (assessments at baseline, 6 months and 12 months)
  Child and caregiver brushing behaviors (11 items) are included in the Basic Research Factors Questionnaire (BRFQ). The BRFQ is a validated questionnaire to assess dental knowledge, attitudes, and behaviors of caregivers with young children. We will also assess frequency of brushing, assistance with brushing, and use of fluoridated toothpaste. The BRFQ is validated in English and has been translated into Spanish (not yet validated) by members of the research team.
Child's dietary intake from the previous day (12:00A - 11:59P) will be captured in-person/telephone/zoom using Nutrition Data System for Research (NDSR) data capture and analysis software | 12 months: from baseline to 12 months post-surgical event. Assessments are at baseline, 6 months and 12 months.
  The software uses interview prompts to conduct a standardized multiple pass 24-hour dietary recall. The multi-pass approach enables respondents to recall foods and beverages consumed with greater accuracy. The parent/caregiver will be asked to use the food amounts booklet to aid the diet interview. A bilingual team member will use the Spanish interviewer prompts provided as an option in the NDSR system for all recalls that are conducted in Spanish. Data collection staff will be trained to conduct dietary recalls. Dietary recall data will be used to calculate nutrient intake (e.g., kcal, fat, protein, carbohydrate) and % kcal from total sugars and added sugars. NDSR is housed on the IHRP network drive which is password protected. Data will be downloaded from the NDSR software package and uploaded to REDCap. The dietary recall interview is validated in both English and Spanish.

SECONDARY OUTCOMES:
The Self-Efficacy Scale for Maternal Oral Care (SESMO) | 12 months: From baseline to 12 months post-surgical event. Assessments are at baseline, 6 months and 12 months.
  The Self-Efficacy Scale for Maternal Oral Care (SESMO) was designed for mothers of children up to 8 years old. It consists of 12 items (on a 4-point Likert scale), divided into two self-efficacy domains (subscales): (i) self-efficacy for tooth brushing and (ii) self-efficacy for dietary habits. This measure has been validated in English and Spanish.
The Multidimensional Assessment of Parenting Scale (MAPS) | 12 months: From baseline to post-surgical event; Assessments are at baseline, 6 months and 12 months.
  The Multidimensional Assessment of Parenting Scale (MAPS) measures parenting practices and includes measures of positive and negative dimensions of warmth/hostility and behavioral control. It includes 34 items on a 5-point Likert scale and has been validated in English and translated into Spanish (not yet validated) by members of the research team.
The Decayed, Missing, Filled Teeth Index (DMFT) | 12 months: From baseline to 12 months post-surgical event at baseline, 6 months and 12 months.
  Clinical Outcomes: The Decayed, Missing, Filled Teeth Index (DMFT) will be used to assess disease severity for primary and any permanent teeth. Scores range from 1-20 if in the primary dentition. Receipt of urgent/emergent dental care or sedation or caries will also be documented. Select members of the research team will extract data from electronic dental records after a child has a preventive dental visit (UIC or MileSquare) and enter into REDCap. We will use this data to calculate the DMFT score, which will be stored in REDCap.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lee, MD, MPH, Principal Investigator — University of Illinois at Chicago
Locations (1):
- College of Dentistry (MC 621), Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: This is our UIC Protect Website. — https://dentistry.uic.edu/protect-research-study/